CLINICAL TRIAL: NCT01107639
Title: Multimodal Therapy With and Without Cetuximab in Patients With Locally Advanced Esophageal Carcinoma - An Open-Label Phase III Trial
Brief Title: Radiation Therapy and Chemotherapy, With or Without Cetuximab, Followed by Surgery in Treating Patients With Locally Advanced Esophageal Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 75/08; 2009-016584-10 (EudraCT Number); EU-21024; CDR0000669249
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2019-05

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Cancer
Keywords: stage IIB esophageal cancer; adenocarcinoma of the esophagus; adenocarcinoma of the gastroesophageal junction; squamous cell carcinoma of the esophagus; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cetuximab; Cisplatin; Docetaxel; Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional immunotherapy (cetuximab) (Experimental): All patients in the experimental arm will be given additional immunotherapy (cetuximab) during cycles 1 and 2, during RT and after surgery.
  Interventions: Biological: cetuximab; Drug: cisplatin; Drug: docetaxel; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy
- Without additional immunotherapy (Active Comparator): Standard therapy without immunotherapy (cetuximab).
  Interventions: Drug: cisplatin; Drug: docetaxel

INTERVENTIONS:
Biological: cetuximab — Loading dose 400 mg/m2 2h infusion Weekly: 250 mg/m2 1h infusion
  Other Names: Erbitux
  Arms: Additional immunotherapy (cetuximab)
Drug: cisplatin — * Cisplatin 75 mg/m2 1h infusion d1, 22
  * Cisplatin 25 mg/m2 1h infusion weekly x5
Drug: docetaxel — * Docetaxel 75 mg/m2 1h infusion d1, 22
  * Docetaxel 20 mg/m2 1/2h infusion weekly x5
  Other Names: Taxotere or generic product
Procedure: adjuvant therapy — During the adjuvant phase, all infusions, given every two weeks, will be at a dose of 500mg/m².
  Arms: Additional immunotherapy (cetuximab)
Procedure: neoadjuvant therapy — During the neoadjuvant phase, the first infusion of cetuximab should be at a dose of 400 mg/m² administered over a period of 2 hours and all subsequent infusions, given weekly, should be of 250 mg/m² over a period of 1 hour, unless any infusion related reaction was observed at a previous infusion. (The maximum infusion rate is 10 mg/min, corresponding to 2 mL/min ready-to-use solution.
  Arms: Additional immunotherapy (cetuximab)

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and to kill tumor cells. Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving radiation therapy together with chemotherapy is more effective with or without cetuximab in treating patients with esophageal cancer.

PURPOSE: This randomized phase III trial is studying giving radiation therapy together with chemotherapy, with or without cetuximab, followed by surgery in treating patients with locally advanced esophageal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of neoadjuvant radiochemotherapy comprising docetaxel, cisplatin, and radiotherapy in combination with cetuximab followed by surgery and adjuvant cetuximab versus neoadjuvant radiochemotherapy comprising docetaxel, cisplatin, and radiotherapy followed by surgery in patients with locally advanced esophageal carcinoma.

Secondary

* To compare the toxicity of the two therapy arms.
* To determine patterns of failure overall and with regard to histology.
* To evaluate economic aspects in a subproject and to perform a radiotherapy quality assurance program.

OUTLINE: This is a multicenter study. Patients are stratified according to center, histology (adenocarcinoma vs squamous cell carcinoma), primary tumor (T2 vs T3-4), and gender (male vs female). Patients are randomized to 1 of 2 treatment arms.

* Arm A:

  * Induction chemotherapy (docetaxel and cisplatin) and concurrent cetuximab Patients receive docetaxel IV over 1 hour and cisplatin IV over 1 hour on day 1 and cetuximab IV over 1-2 hours on day 1, 8, and 15. Treatment repeats every 21 days for 2 courses.
  * Chemotherapy (docetaxel and cisplatin), cetuximab, and concurrent radiotherapy Beginning in week 7, patients receive cetuximab IV over 1 hour, docetaxel IV over 30 minutes, cisplatin IV over 1 hour on days 43, 50, 57, 64, and 71 and undergo radiotherapy 5 days a week for 5 weeks. Patients then undergo surgery 4-7 weeks after completion of radiotherapy.
  * Adjuvant cetuximab Beginning 3-6 weeks after completion of surgery, patients receive cetuximab IV over 1-2 hours once every 2 weeks for a total of 6 doses.
* Arm B: Patients receive induction chemotherapy comprising docetaxel IV and cisplatin IV for 2 courses as in arm A. Beginning in week 7, patients receive docetaxel IV, cisplatin IV, and concurrent radiotherapy for 5 weeks as in arm A. Patients then undergo surgery 4-7 weeks after completion of radiotherapy.

After completion of study therapy, patients are followed up at 1 (arm B) or 6 (arm A) months, every 3 months for 3 years, and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed esophageal carcinoma
* Meets the following criteria:

  * Resectable, locally advanced disease as determined by the combination of CT scan, endoluminal ultrasound (EUS), PET scan, and a multidisciplinary team discussion

    * T2, N1-3; T3, any N; or T4a, any N (if technically resectable with curative intent [R0] as decided by a multidisciplinary team discussion)

      * EUS-guided fine-needle aspiration (FNA) allowed, but determines nodal status only if positive FNA
    * No T1, any N, M0; or T2, N0, M0; T4a (due to infiltration of the trachea-bronchial tree or organ involvement that cannot be operated on with curative intent [R0] as decided by a multidisciplinary team discussion); T4b; or distant metastasis (M1)
  * Type I or II disease according to the Siewert classification
  * Squamous cell carcinoma (including basaloid-squamous cell and adenosquamous carcinoma) or adenocarcinoma of the thoracic esophagus or the esophagogastric junction (from 5 cm below the entrance of the esophagus into the thorax to the gastric cardia)
* Patients with obstructive tumors are eligible (obstructive tumors will be considered as locally advanced tumors)
* No cervical esophageal carcinoma and tumors involving the first 5 cm of the thoracic esophagus
* No airway infiltration in case of tumors at or above the tracheal bifurcation
* No peritoneal carcinomatosis in case of adenocarcinomas infiltrating the gastric cardia (i.e., esophagogastric junction carcinoma Siewert type I or II)

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Creatinine clearance > 60 mL/min
* Bilirubin ≤ 1.0 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* AST ≤ 1.5 times ULN
* INR normal
* PTT ≤ 1.0 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy
* FEV_1 ≥ 1.5 L OR ≥ 75% of the reference value
* Must be compliant and geographically proximal for staging and follow-up
* Considered operable (i.e., appropriate organ functions and ability to undergo general anesthesia)
* No other malignancies within the past 5 years except nonmelanomatous skin cancer or adequately treated carcinoma in situ of the cervix
* No severe or uncontrolled cardiovascular disease, including any of the following:

  * NYHA class III-IV congestive heart failure
  * Unstable angina pectoris
  * Myocardial infarction within the past 12 months
  * Significant arrhythmias
* No psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, and answering questionnaires
* No active uncontrolled infection
* No serious underlying medical condition that, in the opinion of the investigator, could impair the ability of the patient to participate in the trial (e.g., uncontrolled diabetes mellitus or active autoimmune disease)
* No preexisting peripheral neuropathy > grade 1
* No definite contraindications for the use of corticosteroids and antihistamines as premedication
* No known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy to the chest
* At least 30 days since prior treatment in another clinical trial
* No concurrent drugs contraindicated for use with the trial drugs
* No other concurrent anticancer treatments
* No other concurrent experimental drugs or investigational treatments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2010-05-27 (Actual); Primary Completion 2016-10-06 (Actual); Study Completion 2018-12-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | time from randomization to a defined event.
  time from randomization to one of the following events, whichever comes first:
  * Tumor progression at any time (progression of primary tumor or local lymph nodes, appearance of new lesions)
  * Recurrence at local, regional or distant site after surgery
  * Death from any cause

SECONDARY OUTCOMES:
Progression-free survival after surgery | from date of surgery to an event as defined in PFS.
Adverse events according to CTCAE version 4.0 and major postoperative complications | during treatment and follow-up period.
Pathological remission | Assessed according to the tumor regression model of Mandard
Overall survival | time from trial randomization to the date of death from any cause
Time to locoregional failure after R0 resection | from date of surgery to date of first documented loco-regional failure
Time to systemic failure after R0 resection | from date of surgery to date of first documented systemic failure
In-hospital mortality | occurring after surgery but while the patient remains in hospital
Time to progression (TTP) | Time to progression is defined as time from randomization to one of the following events, whichever comes first: - Tumor progression at any time. - Recurrence at local, regional or distant site after surgery. - Death due to tumor

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ruhstaller, MD, Study Chair — Cantonal Hospital of St. Gallen; Michael Stahl, MD, Study Chair — Kliniken Essen-Mitte
Locations (57):
- Austria (7):
  - Landeskrankenhaus, Feldkirch
  - Universitätsklinik für Innere Medizin I, Innsbruck
  - Krankenhaus Barmherzige Schwestern Linz, Linz
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - Universitätsklinikum der PMU Salzburg, Salzburg
  - Universitätsklinik für Innere Medizin, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- France (16):
  - Centre Hospitalier Général, Béziers
  - Hôpital Avicenne, Bobigny
  - Hôtel Dieu Estaing, Clermont-Ferrand
  - Centre Georges-François Leclerc, Dijon
  - CHU Le Bocage, Dijon
  - Centre Bourgogne, Lille
  - CHRU de Lille, Lille
  - Clinique François Chénieux, Limoges
  - CHU la TIMONE, Marseille
  - CH Régional de la Source, Orléans
  - CH Saint Jean, Perpignan
  - Hôpital Haut Leveque, Pessac
  - CHU, Rennes
  - CHU de Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez
  - Clinique Ste Anne, Strasbourg
  - Hôpital Purpan, Toulouse
- Germany (12):
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Kliniken Essen - Mitte, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Klinikum Herford, Herford
  - Klinikum Ludwigsburg, Ludwigsburg
  - Universitaetsklinikum Giessen und Marburg GmbH, Marburg
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Staedtisches Klinikum Solingen, Solingen
  - Klinikum Stuttgart - Katharinenhospital, Stuttgart
  - Universitaetsklinikum Tuebingen, Tübingen
- Szent Laszlo Korhaz, Budapest, Hungary
- Switzerland (21):
  - Hirslanden Klinik Aarau, Aarau
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - St. Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hôpital du Valais (RSV)-CHCVs, Sion
  - Regionalspital, Thun
  - Ospedale Italiano, Viganello
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum Klinik im Park, Zurich
  - Klinik Hirslanden, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruhstaller T, Thuss-Patience P, Hayoz S, Schacher S, Knorrenschild JR, Schnider A, Plasswilm L, Budach W, Eisterer W, Hawle H, Mariette C, Hess V, Mingrone W, Montemurro M, Girschikofsky M, Schmidt SC, Bitzer M, Bedenne L, Brauchli P, Stahl M; Swiss Group for Clinical Cancer Research (SAKK); German Esophageal Cancer Study Group; Austrian 'Arbeitsgemeinschaft Medikamentose Tumortherapie' (AGMT); Federation Francophone de Cancerologie Digestive (FFCD)/Federation de Recherche en Chirurgie (FRENCH). Neoadjuvant chemotherapy followed by chemoradiation and surgery with and without cetuximab in patients with resectable esophageal cancer: a randomized, open-label, phase III trial (SAKK 75/08). Ann Oncol. 2018 Jun 1;29(6):1386-1393. doi: 10.1093/annonc/mdy105. PMID 29635438
- [Derived] von Holzen U, Schmidt S, Hayoz S, Steffen T, Grieder F, Bartsch D, Schnider A, Knoefel WT, Piessen G, Kettelhack C, Marti WR, Schafer M, Fugger R, Koigsrainer A, Gloor B, Furrer M, Gerard MA, Hawle H, Walz MK, Alesina P, Ruhstaller T; Swiss Group for Clinical Cancer Research (SAKK), the German Esophageal Cancer Study Group, the Austrian Arbeitsgemeinschaft Medikamentose Tumortherapie (AGMT), the Federation Francophone de Cancerologie Digestive (FFCD)/Federation de Recherche en Chirurgie (FRENCH). Surgical Outcomes After Neoadjuvant Chemoradiation Followed by Curative Surgery in Patients With Esophageal Cancer: An Intergroup Phase III Trial of the Swiss Group for Clinical Cancer Research (SAKK 75/08). Ann Surg. 2022 Jun 1;275(6):1130-1136. doi: 10.1097/SLA.0000000000004334. Epub 2020 Aug 26. PMID 33055589
- [Derived] Fehr M, Hawle H, Hayoz S, Thuss-Patience P, Schacher S, Riera Knorrenschild J, Durr D, Knoefel WT, Rumpold H, Bitzer M, Zweifel M, Samaras P, Mey U, Kung M, Winterhalder R, Eisterer W, Hess V, Gerard MA, Templeton A, Stahl M, Ruhstaller T; Swiss Group for Clinical Cancer Research (SAKK); German Esophageal Cancer Study Group; Austrian Arbeitsgemeinschaft Medikamentose Tumortherapie (AGMT); Federation Francophone de Cancerologie Digestive (FFCD) / Federation de Recherche en Chirurgie (FRENCH). High thromboembolic event rate in patients with locally advanced oesophageal cancer during neoadjuvant therapy. An exploratory analysis of the prospective, randomised intergroup phase III trial SAKK 75/08. BMC Cancer. 2020 Feb 28;20(1):166. doi: 10.1186/s12885-020-6623-z. PMID 32111181